CLINICAL TRIAL: NCT03914508
Title: An Open Label Pilot Study of Tracking and Behavior Change for Weight Loss in Adults
Brief Title: PACIFIC-FIT: Providing Adults Collaborative Interventions for Ideal Changes Focused Intervention and Tracking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kerri Boutelle, Prinicipal Investigator, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 181514
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Overeating; Body Mass Index; Weight; Treatment; Cravings; Intervention; Behavioral Treatment
MeSH Terms: conditions — Overweight; Obesity; Hyperphagia; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Memory + Behavioral Weight Loss (M+BWL) (Experimental): The M+BWL program will integrate memory interventions to the BWL program. The BWL program will include dietary recommendations, physical activity recommendations, and behavioral change recommendations.
  Interventions: Behavioral: Memory + Behavioral Weight Loss

INTERVENTIONS:
Behavioral: Memory + Behavioral Weight Loss — BWL and memory enhancement (M+BWL) will be integrated to capitalize on the strengths of both treatments. All participants will be taught general behavioral weight loss skills including to decrease caloric intake and increase physical activity, self-monitoring, goal setting, managing high-risk situations, meal planning, slowing eating, problem solving, social support, cognitive restructuring, lapse and relapse prevention skills, and maintaining weight loss. The proposed M+BWL program provides memory interventions based on the literature, including eating attentively, memory of previous meal, memory skills for planning, effects of diet on memory and the relationship between memory and satiety. The M+BWL program will also utilize experiential learning during the group program such as practicing memory enhanced skills during eating.
  Other Names: M+BWL

SUMMARY:
The pilot study will be a one group treatment program and will be utilized to refine the M+BWL program.

DETAILED DESCRIPTION:
The investigators have developed a new model for the treatment of obesity, which emphasizes the role of memory on food consumption in an overweight population.The pilot study will be an open label trial of a memory+behavioral weight loss (M+BWL) group treatment. The treatment will be administered in 14 group sessions over 16 weeks. The investigators will recruit adults with overweight and obesity and will assess them at baseline (prior to treatment), during treatment, post-treatment (immediately following treatment), and follow-up (3 months after treatment). Assessments will include body mass index (BMI), body composition, and binge eating over the course of treatment and follow-up. This study will contribute to the study of basic behavioral mechanisms and food intake, could provide a novel model for the treatment of obesity, and could inform clinical decision making regarding obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be overweight (BMI between 25-45)
2. Participant must be between the ages of 18-65
3. Participant can read at a minimum of an 5th grade level in English
4. Participant is willing to participate and to commit to 16 weeks of treatment and attendance at assessments
5. Participants must consent to audio-taping of assessment interviews and treatment group sessions.
6. Participants will be free of major medical conditions such as a recent history of coronary heart disease; recent history of myocardial infarction; recent symptoms of angina, diabetes, recent stroke, orthopedic problems that would limit activity during the following twelve months; or any other serious medical condition that would make physical activity unsafe.

Exclusion Criteria:

1. Participants will not have bulimia or anorexia, significant cognitive impairment, a known psychotic disorder, or unstable psychiatric illness (e.g., recent psychiatric hospitalization, acute suicidal ideation) as derived from their intake interview and questionnaires.
2. Participants will not be moving out of the San Diego area for the duration of their study enrollment (7 months).
3. Participants will not be pregnant, planning to get pregnant during the 7-month study period or lactating.
4. Participants will not be taking medication for weight loss or that may impair physical activity tolerance or performance.
5. Participants with medical or psychological problems, or taking medications that could make adherence with the study protocol difficult or dangerous, or would influence weight and eating, or cognitive functioning, such as attention, concentration, or mental status will not be included.
6. Participants cannot have a history of bariatric surgery
7. Participants cannot currently be enrolled in an organized weight control program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
body mass index as measured by height and weight | Change from baseline at an average of 4 months and 7 months
  kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, Ph.D., Principal Investigator — UCSD
Locations (1):
- UCSD Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California, United States

REFERENCES:
- [Background] Robinson E, Aveyard P, Daley A, Jolly K, Lewis A, Lycett D, Higgs S. Eating attentively: a systematic review and meta-analysis of the effect of food intake memory and awareness on eating. Am J Clin Nutr. 2013 Apr;97(4):728-42. doi: 10.3945/ajcn.112.045245. Epub 2013 Feb 27. PMID 23446890